CLINICAL TRIAL: NCT02238964
Title: A Randomised Controlled Trial of Reinforcement of Closure of Stoma Site Using a Biological Mesh.
Brief Title: Reinforcement of Closure of Stoma Site
Acronym: ROCSS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: LifeCell (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RG_11-186; 46330337 (Registry Identifier: ISRCTN); 13461 (Registry Identifier: UKCRN); 12/WM/0187 (Other: NRES)
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Strattice™ Reconstructive Tissue Matrix (Active Comparator): Strattice(TM) Reconstructive Tissue Matrix will be placed intra-peritoneally fashion. Once correctly placed, the fascia above will be closed using Prolene, PDS or Nylon (surgeon preference, but excluding Vicryl).
  Interventions: Device: Strattice™ Reconstructive Tissue Matrix
- Standard closure (Active Comparator): Fascial closure will be the preferred technique of the surgeon without mesh reinforcement. The technique recommended is the fascia should be closed with Prolene, PDS or nylon sutures; Vicryl should not be used for the fascia. This technique can include either interrupted or continuous sutures.
  Closure of the muscle, soft tissues and skin is up to the discretion of the operating surgeon.
  Interventions: Procedure: Standard Closure

INTERVENTIONS:
Device: Strattice™ Reconstructive Tissue Matrix — The protocol preference is for the mesh to be placed intra-peritoneally fashion (i.e. below the peritoneum). Anchoring bites will be taken in four to six sites of peritoneum (e.g. using 2-0 PDS) and the mesh will be 'parachuted' into place. Once correctly placed, the fascia above will be closed using Prolene, PDS or Nylon (surgeon preference, but excluding Vicryl). Infiltration of up to 40ml 0.25% Marcaine for infiltration into the fascial layer is recommended. The remainder of the closure will be at the surgeon's discretion.
  Arms: Strattice™ Reconstructive Tissue Matrix
Procedure: Standard Closure — The non-intervention arm for fascial closure will be the preferred technique of the surgeon without mesh reinforcement. The fascia should be closed with Prolene, PDS or nylon sutures; Vicryl should not be used for the fascia. The remainder of the closure will be at the surgeon's discretion.
  Arms: Standard closure

SUMMARY:
ROCSS is a randomised controlled trial of the placement of a biological mesh at the site of stoma closure. Our hypothesis is that reinforcing the stoma closure site with a collagen mesh (Strattice®) is superior to the standard technique in preventing herniation at 2 years.

DETAILED DESCRIPTION:
Closure of complex and contaminated abdominal wounds is challenging and carries risks, including wound dehiscence and incisional hernias. Use of biological meshes in these situations may provide a safe method of reducing these complications, especially long-term incisional hernias. ROCSS will use stoma site closure as a model for biological mesh placement during any difficult contaminated abdominal wall closures.

Hernia at the site of stoma closure occurs in up to 30% of patients and is associated with adverse effects on quality of life. In up to 10% of cases, patients are submitted to complex re-operation which carries significant morbidity. Not all patients will report symptoms or undergo repair, as they do not wish to have a further major operation. Incisional hernias at the site of stomas closure form an important and well defined subgroup. If there is a measurable benefit from mesh insertion, elective use of a collagen mesh would warrant consideration in the closure of other difficult, contaminated abdominal wounds. This study will also provide useful information on the value of using a CT scan as an early diagnostic tool of herniation, which could then be used in future abdominal wall studies as a surrogate endpoint for clinical hernia.

ROCSS aims to assess whether a biological mesh (collagen tissue matrix) reduces the incidence of clinically detectable stoma closure site hernias at two years compared to standard closure techniques. The primary outcome is Occurrence of clinically detectable hernias at two years post randomisation. Other outcomes include surgical re-intervention rate, surgical complications at 30 days post-operation and 1 year post-randomisation, quality of life and post-operative pain, cost-benefit analysis and radiological hernia rate at one year post-randomisation (an exploratory analysis will compare radiological hernia rate at 1 year with clinical hernia rate at 2 years to assess the value of using a CT scan as an early diagnostic tool of incisional hernias).

Randomisation is 1:1 between Strattice® mesh vs. standard closure. The sample size for the trial is 560 (80% power, 10% dropout/crossover, 40% proportional reduction - 25% to 15%) and recruitment will be over 2 years from at least 30 centres. ROCSS will be a double blind (observer blind) randomised controlled trial with a CT scan at one year and clinical follow up at 2 years. Cost benefit analysis and quality of life analysis will be performed at 2 years. The sample size will be reviewed prior to reaching target and may be increased 790 (90% power, 20% dropout/crossover, 40% proportional reduction - 25% to 15%).

ELIGIBILITY:
Inclusion Criteria:

* Require an elective closure of an ileostomy or a colostomy.
* Able and willing to provide written informed consent.
* Aged 18 years or over.

Exclusion Criteria:

* Taking part in another clinical study which is related to the surgical procedure.
* Allergic to any porcine or collagen products.
* History of familial adenomatous polyposis, due to increased risk of desmoid tumours.
* The surgeon determines that a mesh repair will definitely be required e.g. due to large parastomal hernia.
* Unable or unwilling to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 790 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Rate of clinically detectable hernias at two years post-randomisation. | Two years post-randomisation.

SECONDARY OUTCOMES:
Radiological hernia rate at one year post-randomisation. | One year post-randomisation.
  An exploratory analysis will also compare radiological hernia rate at 1 year with clinical hernia rate at 2 years to assess the value of using a CT scan as an early diagnostic tool of incisional hernias.
Incidence of developing a symptomatic hernia evaluated at 12 and 24 months postrandomisation. | One and two years post-randomisation.
  The clinical detection of hernias defined by palpable fascial defects, and global weaknesses around closed stoma sites without palpable fascial defects, will be recorded. Patient-reported hernia symptoms including a local lump or pain at the site of the stoma closure will also be collected.
Surgical re-intervention rates at 2 years post-randomisation. | Two years post-randomisation.
Surgical complications, including wound infections and seroma formation, at 30 days postoperatively and at 1 year post-randomisation. | 30 days postoperatively, 1 year post randomisation
Quality of life assessed using EuroQol EQ-5D at baseline, 30 days post-operatively, 12 and 24 months post-randomisation. | Baseline, 30 days post-operatively, one and two years post-randomisation
Pain assessed using a 100 point visual analogue scale at baseline, 30 days postoperatively, 12 and 24 months post-randomisation. | Baseline, 30 days post-operatively, one and two years post-randomisation
Costs per hernia clinically detected at 2 years post-randomisation. | Two years post-randomisation.
Two-year and long-term costs per additional quality adjusted life (QALY) year gained. | Two-year post-randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Dion G Morton, MD, Principal Investigator — Professor of Colorectal Surgery
Locations (35):
- Hvidovre Hospital, Copenhagen, Denmark
- Academisch Medisch Centrum, Amsterdam, Netherlands
- United Kingdom (33):
  - Tameside General Hospital, Ashton-under-Lyne
  - Royal United Hospital Bath, Bath
  - Heart of England NHS Foundation Trust, Birmingham
  - Queen Elizabeth Hospital, Birmingham
  - Sandwell General Hospital, Birmingham
  - Pilgrim Hospital, Boston
  - Bristol Royal Infirmary, Bristol
  - Broomfield Hospital, Chelmsford
  - St Peters Hospital, Chertsey
  - Chesterfield Royal Hospital, Chesterfield
  - Western Sussex Hospitals NHS Foundation Trust, Chichester
  - University Hospital Coventry, Coventry
  - Doncaster Royal Infirmary, Doncaster
  - Dorset Country Hospital, Dorchester
  - James Paget University Hospital, Great Yarmouth
  - St Marks Hospital, Harrow
  - Raigmore Hospital, Inverness
  - University Hospitals of Leicester NHS Trust, Leicester
  - Macclesfield District General Hospital, Macclesfield
  - Queen Elizabeth the Queen Mother Hospital, Margate
  - Norfolk & Norwich University Hospital, Norwich
  - Queens Medical Centre, Nottingham
  - Salisbury District Hospital, Salisbury
  - University Hospital of North Tees, Stockton-on-Tees
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Kings Mill Hospital, Sutton in Ashfield
  - Manor Hospital, Walsall
  - Royal Albert Edward Infirmary, Wigan
  - New Cross Hosptial, Wolverhampton
  - Worcestershire Royal Hospital, Worcester
  - Wythenshawe Hosptial, Wythenshawe
  - Yeovil District Hospital, Yeovil
  - York Hospital, York

REFERENCES:
- [Derived] Reinforcement of Closure of Stoma Site (ROCSS) Collaborative and West Midlands Research Collaborative. Prophylactic biological mesh reinforcement versus standard closure of stoma site (ROCSS): a multicentre, randomised controlled trial. Lancet. 2020 Feb 8;395(10222):417-426. doi: 10.1016/S0140-6736(19)32637-6. PMID 32035551
- [Derived] Reinforcement of Closure of Stoma Site (ROCSS) Collaborative and the West Midlands Research Collaborative. Feasibility study from a randomized controlled trial of standard closure of a stoma site vs biological mesh reinforcement. Colorectal Dis. 2016 Sep;18(9):889-96. doi: 10.1111/codi.13310. PMID 26924621
- See also: Trial website — http://www.birmingham.ac.uk/ROCSS